CLINICAL TRIAL: NCT02412202
Title: Echocardiographic Detection of Extravascular Lung Water Increase During Weaning From Mechanical Ventilation
Acronym: ECHOBAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DEMOSTHENES MAKRIS, AS. PROFESSOR, University of Thessaly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 273/2015
Record Dates: First submitted 2015-03-27; First posted 2015-04-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Ventilator Weaning

ARMS (1):
- patients who undergo weaning from mechanical ventilation (Other): consecutive mechanically ventilated critical ill patients who fulfil criteria for weaning will be included
  Interventions: Other: Monitoring of pulmonary oedema induced by weaning from mechanical ventilation

INTERVENTIONS:
Other: Monitoring of pulmonary oedema induced by weaning from mechanical ventilation

SUMMARY:
Switching from positive airway pressure ventilation to spontaneous ventilation during weaning from mechanical ventilation, pulmonary edema may occur and in this case, doppler echocardiographic (U/S) indices of cardiac dysfunction correlates with the concentration of fluid in interstitial space.

Forty consecutive mechanically ventilated critical ill patients who fulfill criteria for weaning from mechanical ventilation, will be included in this study. All patients will be evaluated daily and when the patients fulfill weaning criteria them they will undergo a 2-hour spontaneous breathing trial (SBT) through a T-piece.

Before and after SBT cardiopulmonary function will be assessed by thermodilution and echocardiography. In patients with preserved LV systolic function, an echocardiographic index of diastolic dysfunction (E/Em ratio) before preforming SBT may identify high risk patients for increasing extravascular water in weaning.

In addition, the investigators expect to find positive correlations (p<0.05) between pulmonary extravascular lung water and echocardiographic indices (such as E/Em ratio) during SBT.

DETAILED DESCRIPTION:
Pulmonary edema (PE) is an underestimated factor of weaning failure. The interruption of mechanical ventilation

1. increases left ventricular (LV) afterload, sympathetic tone and may provoke myocardial schema, LV dysfunction and
2. augments blood in-flow into the thorax and may cause right ventricular dilation and intraventricular septum left shift.

These events may impair LV compliance during weaning, increase intra-capillary pulmonary pressures and cause cardiogenic PE (CPE). The investigators have recently shown that LV diastolic dysfunction may predispose to weaning failure, while echocardiographic markers of CPE may provide further insight in weaning process. Notably, this could be especially true in chronic obstructive pulmonary disease patients where strategies aiming to manage heart failure (i.e. diuretics, nitroglycerin) has been shown to improve weaning outcomes.

In addition, vigorous inspiratory efforts against the endotracheal tube during spontaneous weaning trials may reduce excessively extracapillary pressures in pulmonary interstitial spaces, causing an intra-pulmonary fluid shift known as negative pressure PE (NPPE).

Primary aim: To study whether echocardiographic parameters of left and right ventricular function, and echocardiographic surrogates of cardiogenic PE (markers of elevated LV filling pressures, such as E/Em) are associated to weaning-induced alterations in extravascular lung water index (EVLWI).

Hypothesis A) Switching from positive airway pressure ventilation to spontaneous ventilation during weaning from mechanical ventilation, pulmonary edema may occur and in this case, doppler echocardiography (U/S) indices of cardiac dysfunction correlates with the concentration of fluid in interstitial space.

B) These events can be further provoked after Maximum Inspiratory Pressure (MIP) trials.

C) Pulmonary edema is a major cause of weaning failure in chronic obstructive pulmonary disease (COPD) patients, even in those without known cardiac disease.

SUBJECTS Thirty-five consecutive mechanically ventilated critical ill patients who fulfil criteria for weaning, will be included.

METHODS All patients will be evaluated daily for the aforementioned weaning criteria and when the patients fulfill them they will undergo A) a 2-hour spontaneous breathing trial (SBT) through a T-piece and B) MIP trial.

Before and after SBT and MIP trials cardiopulmonary function will be assessed by thermodilution and echocardiography.

Extravascular Lung Water Index (EVLWI) study. EVLWI will be assessed by transpulmonary thermodilution (PiCCO plus system, Pulsion Medical Systems and Philips Medical Systems, USA). Transpulmonary thermodilution measures left-side CO by injection of a cold injectate (15-20 ml,10C lower than blood temperature) via subclavian or internal jugular vein and by the detection of the change in temperature in the arterial system via femoral access. Analysis of the thermodilution curve in terms of mean transit time (MTt) and downslope time (DSt) will be used for determination of intra and extra vascular fluid volumes. EVLW correlates to the extravascular thermal volume in the lungs and it is evaluated through the MTt.

Principle parameters obtained by transpulmonary thermodilution are following

* cardiac output (absolute/indexed parameters, CO/CI)
* cardiac function index (CFI)
* extravascular lung water (EVLW/EVLWI)
* pulmonary vascular permeability index (PVPI)
* global ejection fraction (GEF)

Echocardiographic study. Baseline Doppler echocardiographic measurements will be obtained before SBT initiation, while participants will be in pressure support ventilation (pre-SBT). Follow up measurements (end-SBT) in patients who succeeded in the trial, will be collected 120 minutes after SBT initiation. In those participants who fail the procedure, measurements will obtained before reconnection to the ventilator. Doppler echocardiography will be performed as previously described (Philips i33, U.S.A.). Mitral inflow pulsed-wave Doppler signals [peak velocities of early (E) and late (A) LV diastolic filling, E-wave deceleration time (DTE)], Tissue Doppler Imaging(TDI)-derived peak systolic (Sm)/early diastolic (Em)/late diastolic (Am) velocities at the lateral/septal mitral annulus and lateral tricuspid annulus, and color M-mode Doppler velocity of propagation (Vp) will be obtained from the apical 4-chamber view. Analysis will be also performed for "conventional" (E/A ratio) and "advanced" (E/Em, ) echocardiographic indices of LV filling pressures.

Expected Results Recruitment period: three months Analysis of results: three months Based on a previous study contacted by the investigators, echocardiographic variables of LV diastolic dysfunction is expected to be found associated with direct measurements of pulmonary edema (EVLWI). In participants with preserved LV systolic function, an E/Em ratio>7.8 before preforming SBT may identify high risk patients for increasing extravascular water in weaning.

Based on preliminary findings EVLWI values measured in critical patients by the investigators were 2-11 ml/Kg.

The investigators expect to find positive correlations (p<0.05) between EVLWI and E/Em during SBT and MIP trials.

Implications:

The findings of the study will provide further insights in the pathophysiology of weaning. This could be especially true in COPD patients where failure rates are high.

Diagnosis of weaning failure and identification of those patients who are prone to develop LV dysfunction during weaning and weaning outcomes may improve with the application of strategies aiming to manage heart failure (i.e diuretics, nitroglycerin).

EVLW measurements and DE indices will be use as an aid to diagnose and to determine the etiology of pulmonary edema in critical care patients.

These indices may retain the predictive value even in the subset of patients who initially pass SBT; therefore, E/Em pre-SBT could identify patients who will probably fail to remain in SBT.

The relationship between DE indices and EVLWI could be advantageous compared to EVLWI measurement alone, for the quantification of lung edema and the guidance of therapy.

ELIGIBILITY:
Inclusion Criteria:

* adequate oxygenation (pressure of oxygen in arterial blood (PaO2)>60mmHg with fraction of inspired oxygen (FiO2)<40%, PEEP<5-10cmH2O, PaO2/FIO2>150-300)
* stable cardiovascular system (Heart rate<140/min, stable blood pressure, without or very minimal vasopressors)
* absence of sepsis and temperature <38 degree of Celcius
* no respiratory acidosis
* adequate hemoglobin (Hb > 8-10g/dL)
* sufficient (adequate mentation ) arousable Glasgow coma scale >13/15, no continuous sedative infusions
* Ramsay score<3
* stable metabolic status (acceptable levels of electrolytes )
* subjective clinical assessments such as resolution of the acute phase of disease and adequate cough.

Exclusion Criteria:

* atrial fibrillation or other arrhythmias
* insufficiency of tricuspidal valve ( +++),
* continuous venous-venous hemodialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Extravascular water increase during weaning from mechanical ventilation measured by echocardiography and thermodilution method | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Larissa, Larissa, Greece

REFERENCES:
- [Background] Kennedy SK, Weintraub RM, Skillman JJ. Cardiorespiratory and sympathoadrenal responses during weaning from controlled ventilation. Surgery. 1977 Aug;82(2):233-40. PMID 877867
- [Background] Buda AJ, Pinsky MR, Ingels NB Jr, Daughters GT 2nd, Stinson EB, Alderman EL. Effect of intrathoracic pressure on left ventricular performance. N Engl J Med. 1979 Aug 30;301(9):453-9. doi: 10.1056/NEJM197908303010901. PMID 460363
- [Background] Hurford WE, Favorito F. Association of myocardial ischemia with failure to wean from mechanical ventilation. Crit Care Med. 1995 Sep;23(9):1475-80. doi: 10.1097/00003246-199509000-00006. PMID 7664548
- [Background] Boussuges A, Pinet C, Molenat F, Burnet H, Ambrosi P, Badier M, Sainty JM, Orehek J. Left atrial and ventricular filling in chronic obstructive pulmonary disease. An echocardiographic and Doppler study. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):670-5. doi: 10.1164/ajrccm.162.2.9908056. PMID 10934104
- [Background] Routsi C, Stanopoulos I, Zakynthinos E, Politis P, Papas V, Zervakis D, Zakynthinos S. Nitroglycerin can facilitate weaning of difficult-to-wean chronic obstructive pulmonary disease patients: a prospective interventional non-randomized study. Crit Care. 2010;14(6):R204. doi: 10.1186/cc9326. Epub 2010 Nov 15. PMID 21078149
- [Background] Isakow W, Schuster DP. Extravascular lung water measurements and hemodynamic monitoring in the critically ill: bedside alternatives to the pulmonary artery catheter. Am J Physiol Lung Cell Mol Physiol. 2006 Dec;291(6):L1118-31. doi: 10.1152/ajplung.00277.2006. Epub 2006 Aug 4. PMID 16891389